CLINICAL TRIAL: NCT05248997
Title: A Phase 2/3, Double-Blind, Randomized, Placebo-Controlled, Safety and Efficacy Trial of BHV-3000 (Rimegepant) Orally Disintegrating Tablet (ODT) for the Acute Treatment of Chronic Rhinosinusitis (CRS) With or Without Nasal Polyps
Brief Title: Safety and Efficacy of BHV-3000 (Rimegepant) Orally Disintegrating Tablet for the Acute Treatment of Chronic Rhinosinusitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHV3000-316; C4951015 (Other: Alias Study Number)
Record Dates: First submitted 2022-01-31; First posted 2022-02-21 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Chronic Rhinosinusitis (CRS) With and Without Nasal Polyps
Keywords: Chronic Rhinosinusitis (CRS); Chronic Rhinosinusitis (CRS) with Nasal Polyps; Chronic Rhinosinusitis (CRS) without Nasal Polyps
MeSH Terms: interventions — rimegepant sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- rimegepant 75 mg ODT (Active Comparator): One dose of rimegepant 75 mg ODT
  Interventions: Drug: rimegepant 75 mg ODT
- Matching Placebo (Active Comparator): One dose of matching placebo
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: rimegepant 75 mg ODT — One dose of rimegepant 75 mg ODT
  Arms: rimegepant 75 mg ODT
Drug: Matching placebo — One dose of matching placebo
  Arms: Matching Placebo

SUMMARY:
The purpose of this study is to compare the efficacy and safety of rimegepant versus placebo in the acute treatment of chronic rhinosinusitis (CRS) with and without nasal polyps.

ELIGIBILITY:
Inclusion Criteria:

* At least two episodes of facial pain/pressure/fullness of moderate or severe intensity on a 4-point rating scale (0 = None, 1 = Mild, 2 = Moderate, 3 = Severe) in the past 30 days prior to the Screening Visit.
* Subject agrees to study-required medication restrictions and the restriction of not starting new medication to treat CRS symptoms during the course of the study.
* Subject agrees to study-required birth control methods during the course of the study, and female subjects must not be breastfeeding.
* No clinically significant abnormality identified on the medical or laboratory evaluation.

Exclusion Criteria:

* Subject has primary headache disorder.
* Subject has history of nasal or facial surgery within the 6 months prior to screening.
* Subject has ongoing rhinitis medicamentosa.
* Subject has diagnosed or suspected invasive fungal rhinosinusitis.
* Subject is currently receiving aspirin desensitization or maintenance therapy for Samter's Triad.
* Subject has a history of recurrent acute sinusitis (four or more episodes per year of acute bacterial rhinosinusitis (ABRS) without signs or symptoms of rhinosinusitis between episodes).
* Body Mass Index > 35.0kg/m2
* Subject history of exclusionary medical conditions such as HIV disease, cardiovascular conditions, uncontrolled hypertension or diabetes, psychiatric conditions, drug or alcohol abuse, malignancies, drug allergies, or any significant and/or unstable medical conditions.
* Subjects taking/using excluded therapies.
* Participation in clinical trial with non-biological investigational agents or investigational interventional treatments.
* Subjects who have previously participated in any BHV-3000/ BMS-927711/ rimegepant study.
* Planned participation in any other investigational clinical trial while participating in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (33):
- United States (33):
  - San Diego Clinical Research Center, La Mesa, California
  - Velocity Clinical San Diego, La Mesa, California
  - National Research Institute, Panorama City, California
  - Sacramento Ear Nose and Throat Surgical and Medical Group, Inc., Roseville, California
  - Sharp & Children's MRI Center, LLC (CT scan), San Diego, California
  - Breathe Clear Institute, Torrance, California
  - Colorado ENT & Allergy, Colorado Springs, Colorado
  - Velocity Clinical Research, New Smyrna Beach, Edgewater, Florida
  - The Medici Medical Research, LLC, Hollywood, Florida
  - Avantis Clinical Research, Miami, Florida
  - Clinovation Research, Pompano Beach, Florida
  - Treasure Valley Medical Research, Boise, Idaho
  - ChicagoENT, Chicago, Illinois
  - Kentuckiana Ear, Nose & Throat, Louisville, Kentucky
  - Best Clinical Trials, LLC (Administrative Only), New Orleans, Louisiana
  - George Stanley Walker, MD, New Orleans, Louisiana
  - University of Missouri Hospital & Clinics, ENT & Allergy Center of Missouri, Columbia, Missouri
  - University of Missouri Healthcare - Investigational Pharmacy, Columbia, Missouri
  - University of Missouri Hospital (Radiology), Columbia, Missouri
  - Clinvest Research, LLC, Springfield, Missouri
  - St Charles Clinical Research, Weldon Spring, Missouri
  - Northwell Health Department of Otolaryngology, New Hyde Park, New York
  - Tekton Research, Inc., Edmond, Oklahoma
  - Allergy, Asthma & Clinical Research Center, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - Velocity Clinical Research, Grants Pass, Grants Pass, Oregon
  - Velocity Clinical Research, Medford, Medford, Oregon
  - Velocity Clinical Research, Anderson, Anderson, South Carolina
  - Carolina ENT Clinic/CENTRI Inc., Orangeburg, South Carolina
  - Spokane Ear, Nose & Throat/ Columbia Surgical Specialists, Spokane, Washington
  - Principle Research Solutions, Spokane, Washington
  - Spokane Ear, Nose & Throat / Columbia Surgical Specialists, Spokane, Washington
  - Allergy, Asthma & Sinus Center, S.C., Greenfield, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=BHV3000-316

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 261 participants were enrolled and randomized in the study. Amongst which 99 received rimegepant and 105 received placebo.
Pre-assignment Details: Participants were to administer one dose of study medication only when participant had a facial pain/pressure/fullness that reached intensity of greater than or equal to (>=) 6 on the numeric rating scale (NRS, 0 to 10) and they had completed pre-dose assessments in electronic (e)-diary. Study medication was to be administered only within 45 days of randomization.
Groups:
- Rimegepant 75 mg: Participants were randomized for administration of rimegepant 75 mg, single dose, orally, as an orally disintegrating tablet (ODT) sublingually.
- Placebo: Participants were randomized for administration of placebo (matched to rimegepant), single dose, orally, as an ODT sublingually.
Period: Overall Study
Arm/Group | Rimegepant 75 mg | Placebo
Started | 131 | 130
Treated | 99 | 105
Completed | 98 | 104
Not Completed | 33 | 26
Not completed — Lost to Follow-up | 1 | 1
Not completed — Randomized but not treated | 32 | 25

BASELINE CHARACTERISTICS:
Groups:
- Rimegepant 75 mg: Participants were randomized for administration of rimegepant 75 mg, single dose, orally, as an ODT sublingually.
- Total: Total of all reporting groups
Arm/Group | Rimegepant 75 mg | Placebo | Total
Number analyzed (Participants) | 131 | 130 | 261
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.6 (15.27) | 49.9 (15.83) | 49.3 (15.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 68 | 145
  Male | 54 | 62 | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 36 | 63
  Not Hispanic or Latino | 102 | 93 | 195
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 19 | 17 | 36
  White | 106 | 105 | 211
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Facial Pain/Pressure/Fullness on NRS at 2 Hours Post-Dose
Description: Facial pain/pressure/fullness was assessed using an NRS score ranging in integers from 0 to 10, with 0 being "no facial pain/pressure/fullness" and 10 being "worst imaginable facial pain/pressure/fullness." Higher scores signified worse condition.
Time Frame: Baseline, 2 hours post-dose
Population: Modified Intent to Treat (mITT) analysis set included randomized participants that received study therapy, had a facial pain/pressure/fullness which reached pain intensity of >= 6 on the NRS (0-10) prior to administration of treatment and provided at least one post-baseline efficacy data point in the e-diary. All assessments after rescue medication administration were set to missing. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 89 | 92
Scores on a scale | -2.70 [-3.16 to -2.25] | -2.61 [-3.06 to -2.17]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p = 0.7782, Linear model (LM) — LM included baseline value as covariate,& fixed effects for treatment group,stratification factor,scheduled time point(TP),TP by treatment group interaction.Repeated measures:modelled by unstructured covariance structure for within participant error; Difference in least square mean = -0.09, 95% CI 2-sided [-0.71 to 0.53]

2. Secondary Outcome: Change From Baseline in Total Nasal Symptom Score (TNSS) at 2 Hours Post-Dose
Description: TNSS was calculated as the sum of 3 symptom scores: facial pain/pressure/fullness, score ranged from 0 (no facial pain/pressure/fullness) to 10 (worst imaginable facial pain/pressure/fullness); nasal obstruction (congestion), score ranged from 0 (no nasal obstruction (congestion) to 10 (worst imaginable nasal obstruction (congestion); and nasal discharge, score ranged from 0 (no nasal discharge) to 10 (worst nasal discharge). TNSS overall score ranged from 0 (no nasal symptom) to 30 (worst nasal symptom); higher scores signified worse condition.
Time Frame: Baseline, 2 hours post-dose
Population: mITT analysis set included randomized participants that received study therapy, had a facial pain/pressure/fullness which reached pain intensity of >= 6 on the NRS (0-10) prior to administration of treatment and provided at least one post-baseline efficacy data point in the e-diary. All assessments after rescue medication administration were set to missing. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 89 | 92
Scores on a scale | -7.04 [-8.16 to -5.91] | -6.74 [-7.85 to -5.64]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p = 0.7079, Linear model (LM) — LM included baseline value as covariate, and fixed effects for treatment group,stratification factor,scheduled TP, TP by treatment group interaction.Repeated measures:modelled by unstructured covariance structure for within participant error; Difference in least square mean = -0.29, 95% CI 2-sided [-1.83 to 1.24]

3. Secondary Outcome: Change From Baseline in Nasal Obstruction (Congestion) at 2 Hours Post-Dose
Description: Nasal obstruction (congestion) severity was assessed using a NRS ranging in integers from 0 (no nasal obstruction [congestion]) to 10 (worst imaginable nasal obstruction [congestion]). Higher scores signified worse condition.
Time Frame: Baseline, 2 hours post-dose
Population: mITT analysis set included randomized participants that received study therapy, had a facial pain/pressure/fullness which reached pain intensity of >=6 on the NRS (0-10) prior to administration of treatment and provide at least one post-baseline efficacy data point in the e-diary. All assessments after rescue medication administration were set to missing. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 89 | 92
Scores on a scale | -2.48 [-2.91 to -2.05] | -2.25 [-2.67 to -1.82]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p = 0.4398, Linear model (LM) — [p-value comment as in outcome 2, analysis 1]; Difference in least square mean = -0.23, 95% CI 2-sided [-0.81 to 0.36]

4. Secondary Outcome: Change From Baseline in Nasal Discharge at 2 Hours Post-Dose
Description: Nasal discharge severity was assessed using a NRS ranging in integers from 0 (no nasal discharge) to 10 (worst imaginable nasal discharge). Higher scores signified worse condition.
Time Frame: Baseline, 2 hours post-dose
Population: mITT analysis set included randomized participants that received study therapy, had a facial pain/pressure/fullness which reached pain intensity of >= 6 on the NRS (0-10) prior to administration of treatment and provide at least one post-baseline efficacy data point in the e-diary. All assessments after rescue medication administration were set to missing. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 89 | 92
Scores on a scale | -1.81 [-2.22 to -1.41] | -1.85 [-2.25 to -1.45]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p = 0.8890, Linear model (LM) — [p-value comment as in outcome 2, analysis 1]; Difference in least square mean = 0.04, 95% CI 2-sided [-0.51 to 0.59]

5. Secondary Outcome: Percentage of Participants With Headache Pain Relief at 2 Hours Post-Dose
Description: Headache pain relief was defined as a headache pain level of none or mild at 2 hours post-dose on a 4-point Likert scale (0 = None; 1 = Mild; 2 = Moderate; 3 = Severe).
Time Frame: 2 hours post-dose
Population: mITT analysis set analyzed. Participants who reported a headache pain level of moderate or severe intensity at baseline were assessed. Participants who had missing data at 2 hours post-dose, or who took rescue medication at or before 2 hours post-dose were imputed as failures. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 69 | 81
Percentage of Participants | 59.4 [47.8 to 71.0] | 55.6 [44.7 to 66.4]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p = 0.6412, Mantel-Haenszel; Stratified by presence of nasal polyps at randomization with Mantel-Haenszel risk estimation; Percentage difference = 3.8, 95% CI 2-sided [-12.1 to 19.7]

6. Secondary Outcome: Percentage of Participants Who Used Rescue Medication Within 24 Hours Post-dose
Description: Post 2 hours after dosing with study medication and after the 2-hour assessments were completed on the e-diary, participants were permitted to use the following rescue medications (non-study medications) such as: acetaminophen or aspirin, ibuprofen, naproxen (or any other type of nonsteroidal anti-inflammatory drug [NSAID]), oral antihistamines (non- sedating), oral decongestants, topical nasal decongestants, topical nasal anticholinergics.
Time Frame: Through 24 hours post-dose
Population: mITT analysis set included randomized participants that received study therapy, had a facial pain/pressure/fullness which reached pain intensity of greater than or equal to (>=) 6 on the NRS (0-10) prior to administration of treatment and provided at least one post-baseline efficacy data point in the e-diary. Participants who recorded rescue medication use within 24 hours post-dose were considered failures, where failure was the event being analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 96 | 100
Percentage of Participants | 7.3 [2.1 to 12.5] | 10.0 [4.1 to 15.9]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p = 0.5001, Mantel-Haenszel; Stratified by presence of nasal polyps at randomization with Mantel-Haenszel risk estimation; Percentage difference = -2.7, 95% CI 2-sided [-10.6 to 5.2]

ADVERSE EVENTS:
Time Frame: Within 7 (+2) days post single administration of study medication (single dose was to be administered on any day from randomization to 45 days post randomization)
Description: Safety analysis set was evaluated.
Groups:
- Rimegepant: Participants received one dose of Rimegepant at a dose of 75 mg, orally, as an ODT for the acute treatment of CRS with or without nasal polyps.
- Placebo: Participants received one dose of Rimegepant matching placebo, orally, as an ODT for the acute treatment of CRS with or without nasal polyps.
Arm/Group | Rimegepant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/105
Other Adverse Events (participants affected / at risk) | 4/99 | 5/105
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rimegepant (N=99) | Placebo (N=105)
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Electrocardiogram PR shortened (Investigations) | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT05248997/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-14): https://cdn.clinicaltrials.gov/large-docs/97/NCT05248997/SAP_001.pdf